CLINICAL TRIAL: NCT02918383
Title: Differential Subchondral Perfusion Mapping Using Indocyanin Green Laser Angiography
Brief Title: Subchondral Perfusion Mapping Using Indocyanin Green Laser
Acronym: ICG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has decided to close the study.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Lee Zuckerman, MD, Assistant Professor, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5160045
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Distal Femoral; Proximal Tibial; Knee Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanin Green Dye (ICG) (Other): Once the patient is in the operating room, the operative intervention will take proceed as current standard protocol dictates for the described procedure. No changes in operative technique will be undertaken apart from injection of the dye and visualization with the camera. After the articular surface of the distal femur or proximal tibia has been exposed, 2.5 mg of indocyanin green will be injected intravenously by anesthetist through a pre-existing IV line outside the sterile field. The operating surgeon will grade 6 locations on a standard scale of chondromalacia or cartilage damage.
  Interventions: Diagnostic Test: Indocyanin Green Dye (ICG)

INTERVENTIONS:
Diagnostic Test: Indocyanin Green Dye (ICG)

SUMMARY:
Laser Angiography using indocyanin green (ICG) is a relatively new technique and has been utilized to assess the viability of soft tissue, most prominently in the general surgery and plastic surgery literature. This technique has been used for prediction of soft tissue viability by assessing the perfusion status. There is currently no Orthopaedic literature regarding the use of this device for assessment of subchondral perfusion of articular surfaces such as the distal femur or other chondral surfaces.

In this pilot study, the use of ICG to detect the perfusion status of a distal femur and proximal tibia during a surgical approach to the knee and correlating this to visible signs of arthritis. For example, due to the difference visible with ICG angiography correlate to gross changes in the cartilage health visible to the naked eye with radiographic imaging.

DETAILED DESCRIPTION:
ICG has been FDA registered since 1959 and is a negatively charged, water-soluble, tricarbocyanine. It binds readily to plasma proteins after injection with almost exclusive bile excretion, and possesses an extremely low toxicity profile. In plasma, ICG has an absorption peak around 807 nm and an emission peak around 822 nm, both within the infrared range. ICG has a short half-life of 150-180 seconds, making multiple administrations possible intra-operatively. It is given intravenously during administration1-4. After it is given through an IV, it is rapidly distributed throughout the circulatory system. When a light of a specific wavelength interacts with the dye, the dye fluoresces in the near-infrared range, which can be acquired by a special camera.

In daily practice, both visualization and palpation are used to provide information about the health of articular cartilage, be it through arthroscopy or open treatment. However, real time assessment of cartilage viability and subchondral perfusion has not been available. Determination of the perfusion status of cartilage surfaces via intra-operative modalities may provide valuable information diagnostically, as well as guide therapeutic intervention. Some possible uses for this technology may be diagnosing and treating osteochondral defects, predicting future osteoarthritis, delineating or predicting areas of avascular necrosis, or use in oncologic surgery. It is currently thought that because this dye currently works extremely well in the soft tissue literature, this will directly translate to being able to accurately assess subchondral bone perfusion.

The incidence of symptomatic knee arthritis in the United States approaches 50% of the population by the time the patient turns 85 and has been shown to significantly impact a patient's quality of life. In 2003, the United States spent $128 billion on arthritis expenditures. Arthritis can be described as the degeneration, or absence of, healthy cartilage. The current way to intra-operatively assess cartilage viability is through inspection and palpation, although this is obviously not always indicative of the overall health of the cartilage. Although an MRI may be obtained pre-operatively showing similar information, this is costly and does not provide the same information that can be assessed intra-operatively. Furthermore, an MRI does not provide information on the perfusion status of the cartilage.

It is our belief that this imaging modality will provide valuable information diagnostically and be able to guide surgical decision making regarding treatments for patients. For example, prior to undergoing a unicompartmental knee replacement, if a patient is found to have degenerative changes of the other compartments, the surgeon may convert to a total knee arthroplasty. If a patient has an osteochondral defect, knowing the perfusion status may provide information on whether to reconstruct the defect with an allograft or drill the defect. A patient undergoing a cruciate retaining total knee arthroplasty may benefit from knowing if the posterior cruciate ligament is pathologic, leading to a posterior stabilized knee replacement. For a patient with avascular necrosis, valuable prognostic information on the viability of their cartilage may help determine if joint preserving surgery is possible. The use of intra-operative ICG may have an impact on intra-operative decision making as the perfusion observed may predict the overall health of structures we currently have no way of assessing in real-time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective orthopedic intervention in which the distal femoral or proximal tibial articular surface is visualized through arthroscopic or open technique
* Patients not meeting exclusion criteria

Exclusion Criteria:

* Iodine allergy
* Intolerance to indocyanine green dye
* Active infection at surgical site
* Known pregnancy
* Inability to comprehend consent process
* Age <18 or > 89
* Significant blood loss risk without tourniquet inflation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Differential Subchondral Perfusion Mapping using Indocyanin Green Laser Angiography | 15 months
  Visible grade of chondromalacia from the 6 points mentioned above.
  * Video will be acquired using the Spy Elite or Pinpoint system of the distal femur or proximal tibial surface. Currently, the software with the SPY elite is able to quantify the degree of dye uptake, and this dye uptake number from the 6 points will also be recorded.
  * Video data will be given a key that corresponds to the subject, thus no videos will be labelled with patient data or information chondromalacia ondromalacia from the 6 points mentioned above.
  * Video will be acquired using the Spy Elite or Pinpoint system of the distal femur or proximal tibial surface. Currently, the software with the SPY elite is able to quantify the degree of dye uptake, and this dye uptake number from the 6 points will also be recorded.
  * Video data will be given a key that corresponds to the subject, thus no videos will be labelled with patient data or information

CONTACTS AND LOCATIONS:
Overall Officials: Lee Zuckerman, MD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Healthcare Department of Orthopaedic Surgery, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No